CLINICAL TRIAL: NCT00021671
Title: Phase III Trial of Antibiotics to Reduce Chorioamnionitis-Related Perinatal HIV Transmission
Brief Title: Antibiotics to Reduce Chorioamnionitis-Related Perinatal HIV Transmission
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: HIVNET 024; 11622 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2001-07-31; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Ampicillin; Nevirapine; Disease Transmission, Vertical; Anti-Infective Agents; Erythromycin; Reverse Transcriptase Inhibitors; Metronidazole; Anti-HIV Agents; Chorioamnionitis; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Chorioamnionitis | interventions — Erythromycin; Nevirapine; Ampicillin; Metronidazole

INTERVENTIONS:
Drug: Erythromycin
Drug: Nevirapine
Drug: Ampicillin sodium
Drug: Metronidazole

SUMMARY:
The purpose of this study is to see if antibiotic drugs given to treat an infection of the uterus during pregnancy can reduce the chances of HIV being passed from an HIV-positive mother to her baby.

A link between bacterial disease of the vagina, premature birth, infection of the uterus during pregnancy, and the passing of HIV from a mother to her baby has been found. Early treatment of these problems may reduce the risk of passing HIV from an HIV-positive mother to her baby.

[Note: As of 02/21/03, enrollment into this study was halted because preliminary data showed that the study antibiotics were not effective in preventing mother-to-child HIV transmission.]

DETAILED DESCRIPTION:
Obstetric risk factors for HIV maternal-child transmission (MCT) include preterm birth, prolonged rupture of the membranes, and chorioamnionitis. Many preterm births are associated with and likely caused by chorioamnionitis. The relationship between bacterial vaginosis, preterm birth, histologic chorioamnionitis, and perinatal transmission of HIV has been consistently demonstrated. Perinatal HIV transmission is more common in preterm infants, and there is now evidence that subclinical chorioamnionitis is a substantial risk factor for MCT. For this study, the primary hypothesis is that early and appropriate treatment of subclinical chorioamnionitis prior to the onset of spontaneous preterm labor, and/or antibiotic treatment during labor, to prevent premature rupture of membrane-associated-chorioamnionitis, will reduce the risk of perinatal HIV transmission.

[Note: As of 02/21/03, enrollment into this study was halted because preliminary data showed that the study antibiotics were not effective in preventing mother-to-child HIV transmission.]

At 20 to 24 weeks, women who are randomized to receive antibiotics receive metronidazole and erythromycin for 7 days. Women randomized to the control group receive identically appearing placebos. With the onset of contractions and/or premature rupture of membranes, study participants will initiate a second oral course of antibiotics consisting of metronidazole and ampicillin or placebo every 4 hours, continuing after delivery until the course is completed. All HIV-infected women and their neonates will be offered the HIVNET 012 nevirapine (NVP) regimen. If the mother accepts the NVP for herself and her baby, she will be given 1 dose of NVP to be taken at onset of labor, and her baby will receive 1 dose of NVP at 72 hours post-birth or discharge, whichever occurs earlier. If the mother refuses NVP or is uninfected, she will receive a matched placebo at the 26- to 30-week visit to preserve participant confidentiality. This study takes place in Blantyre and Lilongwe, Malawi, in Lusaka, Zambia, and in Dar es Salaam, Tanzania.

ELIGIBILITY:
Inclusion Criteria

* HIV positive.
* 20 to 24 weeks pregnant.
* Willing to take the planned antibiotic treatment.
* Planning to deliver at 1 of the study sites.
* Willing to come back for follow-up visits for 1 year after the baby is born.

Exclusion Criteria

* Have taken antibiotics, except for syphilis or gonorrhea, within the last 2 weeks.
* Are allergic to penicillin, ampicillin, erythromycin, or metronidazole.
* Have major illnesses, such as diabetes, severe kidney or heart disease, or active tuberculosis, which might affect the pregnancy.
* Are having major problems with the pregnancy, such as placenta previa, ruptured membranes, or multiple pregnancy.
* Have a central nervous system disease, such as seizures.
* Are taking anticoagulant drugs.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3720
Dates: Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taha E Taha, MD, PhD, Study Chair — Johns Hopkins University; Robert Goldenberg, MD, Study Chair — Department of Obstetrics and Gynecology, University of Alabama at Birmingham
Locations (1):
- Megan Valentine, Research Triangle Park, North Carolina, United States

REFERENCES:
- [Background] Goldenberg RL, Andrews WW, Yuan AC, MacKay HT, St Louis ME. Sexually transmitted diseases and adverse outcomes of pregnancy. Clin Perinatol. 1997 Mar;24(1):23-41. PMID 9099500
- [Background] St Louis ME, Kamenga M, Brown C, Nelson AM, Manzila T, Batter V, Behets F, Kabagabo U, Ryder RW, Oxtoby M, et al. Risk for perinatal HIV-1 transmission according to maternal immunologic, virologic, and placental factors. JAMA. 1993 Jun 9;269(22):2853-9. PMID 8098783
- [Background] Hauth JC, Goldenberg RL, Andrews WW, DuBard MB, Copper RL. Reduced incidence of preterm delivery with metronidazole and erythromycin in women with bacterial vaginosis. N Engl J Med. 1995 Dec 28;333(26):1732-6. doi: 10.1056/NEJM199512283332603. PMID 7491136
- [Background] Mercer BM, Miodovnik M, Thurnau GR, Goldenberg RL, Das AF, Ramsey RD, Rabello YA, Meis PJ, Moawad AH, Iams JD, Van Dorsten JP, Paul RH, Bottoms SF, Merenstein G, Thom EA, Roberts JM, McNellis D. Antibiotic therapy for reduction of infant morbidity after preterm premature rupture of the membranes. A randomized controlled trial. National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. JAMA. 1997 Sep 24;278(12):989-95. PMID 9307346
- [Result] Chi BH, Wang L, Read JS, Sheriff M, Fiscus S, Brown ER, Taha TE, Valentine M, Goldenberg R. Timing of maternal and neonatal dosing of nevirapine and the risk of mother-to-child transmission of HIV-1: HIVNET 024. AIDS. 2005 Nov 4;19(16):1857-64. doi: 10.1097/01.aids.0000189863.82429.2f. PMID 16227794
- [Result] Goldenberg RL, Mudenda V, Read JS, Brown ER, Sinkala M, Kamiza S, Martinson F, Kaaya E, Hoffman I, Fawzi W, Valentine M, Taha TE; HPTN 024 Study Team. HPTN 024 study: histologic chorioamnionitis, antibiotics and adverse infant outcomes in a predominantly HIV-1-infected African population. Am J Obstet Gynecol. 2006 Oct;195(4):1065-74. doi: 10.1016/j.ajog.2006.05.046. Epub 2006 Jul 26. PMID 16875654
- [Result] Goldenberg RL, Mwatha A, Read JS, Adeniyi-Jones S, Sinkala M, Msmanga G, Martinson F, Hoffman I, Fawzi W, Valentine M, Emel L, Brown E, Mudenda V, Taha TE; Hptn024 Team. The HPTN 024 Study: the efficacy of antibiotics to prevent chorioamnionitis and preterm birth. Am J Obstet Gynecol. 2006 Mar;194(3):650-61. doi: 10.1016/j.ajog.2006.01.004. PMID 16522393
- [Derived] Mwinga K, Vermund SH, Chen YQ, Mwatha A, Read JS, Urassa W, Carpenetti N, Valentine M, Goldenberg RL. Selected hematologic and biochemical measurements in African HIV-infected and uninfected pregnant women and their infants: the HIV Prevention Trials Network 024 protocol. BMC Pediatr. 2009 Aug 7;9:49. doi: 10.1186/1471-2431-9-49. PMID 19664210
- [Derived] Chi BH, Wang L, Read JS, Taha TE, Sinkala M, Brown ER, Valentine M, Martinson F, Goldenberg RL. Predictors of stillbirth in sub-saharan Africa. Obstet Gynecol. 2007 Nov;110(5):989-97. doi: 10.1097/01.AOG.0000281667.35113.a5. PMID 17978109
- [Derived] Goldenberg RL, Andrews WW, Hoffman I, Fawzi W, Valentine M, Young A, Read JS, Brown ER, Mudenda V, Kafulafula G, Mwinga K, Taha TE. Fetal fibronectin and adverse infant outcomes in a predominantly human immunodeficiency virus-infected African population: a randomized controlled trial. Obstet Gynecol. 2007 Feb;109(2 Pt 1):392-401. doi: 10.1097/01.AOG.0000247628.68415.00. PMID 17267841